CLINICAL TRIAL: NCT00185770
Title: Reducing Television Viewing to Prevent Childhood Obesity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL062224 (NIH); R01HL062224 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Obesity; Cardiovascular Diseases
Keywords: Obesity prevention; Television; Screen time; Schools; Preadolescents
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Reducing television and other screen time (SMART curriculum)

SUMMARY:
Randomized controlled trial to test the efficacy of reducing television, videotape and video game use to prevent obesity, increase physical activity, improve physical fitness, and decrease dietary fat and calorie intake among third grade children in twelve ethnically-diverse elementary schools.

DETAILED DESCRIPTION:
The United States has experienced dramatic increases in obesity among both children and adults. Population-based primary prevention may hold the greatest promise. Unfortunately, obesity prevention programs that have specifically attempted to reduce fat and calorie intake and increase physical activity have been relatively ineffective at reducing body fatness. As a result, there is a pressing need for innovative interventions to prevent obesity.

Children spend more time watching television and videotapes and playing video games than in any other activity except sleeping. As a result, there has been widespread speculation that television viewing might be one of the most easily modifiable causes of obesity among children. This hypothesis has broad appeal, but has been difficult to validate. Epidemiological studies have consistently found weak associations between media use and childhood obesity, and additional epidemiological studies are unlikely to help clarify these relationships.

We propose an innovative experimental model. In the current environment, in which television viewing is already so prevalent, the question of greatest clinical, practical and policy importance is: Will reducing television, videotape and video game use prevent childhood obesity? As a foundation for this proposal, we have completed two pilot studies that demonstrate (1) it is possible to significantly reduce children's television, videotape and video game use and (2) that a school-based intervention to reduce children's television, videotape and video game use may result in clinically significant decreases in adiposity.

We propose a school-based randomized controlled trial involving 12 ethnically- and socioeconomically-diverse elementary schools and approximately 900 third graders. Six schools will be randomly assigned to receive an intervention to reduce television, videotape and video game use and the other six schools will receive an attention-placebo control intervention, to minimize the potential for compensatory rivalry or resentful demoralization. Our proposed intervention model is derived directly from principles of Bandura's social cognitive theory and includes a classroom curriculum and parent newsletters. The primary intervention will be delivered throughout the third grade school year.

Survey and physical assessments of all children will occur at baseline, at the end of 3rd grade (post-test) and at the beginning and end of 4th grade (4 month and one year follow-ups, respectively). A subsample of children will participate in 4 days of activity monitoring and three 24-hour dietary recalls at baseline, post-test and one-year follow-up. Parents will be interviewed by phone.

PRIMARY HYPOTHESIS: Compared to controls, third grade children exposed to a school-based intervention to reduce time spent watching television and videotapes and playing video games, will significantly reduce their body mass index (BMI, kg/m2). In addition, triceps skinfold thickness and waist and hip ratio will be measured to further characterize changes in obesity resulting from the intervention.

SECONDARY HYPOTHESES: Children attending intervention schools will significantly decrease the amount of time they spend watching television, watching videotapes and playing video games; Children attending intervention schools will significantly increase their levels of moderate to vigorous physical activity and total physical activity; Children attending intervention schools will significantly improve their physical fitness; Children attending intervention schools will significantly reduce their fat intakes and total calorie intakes; Children attending intervention schools will significantly reduce the number of meals and snacks they eat while watching television and videotapes or playing video games.

ELIGIBILITY:
Inclusion Criteria:

* All 3rd grade students attending the participating elementary schools.

Exclusion Criteria:

* Unable to complete the study procedures

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 1999-04

PRIMARY OUTCOMES:
body mass index

SECONDARY OUTCOMES:
prevalence/incidence of obesity
triceps skinfold thickness
waist circumference
screen time
physical activity
cardiorespiratory fitness
dietary intake
weight concerns
academic performance

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N. Robinson, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Robinson TN. Television viewing and childhood obesity. Pediatr Clin North Am. 2001 Aug;48(4):1017-25. doi: 10.1016/s0031-3955(05)70354-0. PMID 11494635
- [Background] Robinson TN. Population-based obesity prevention for children and adolescents. In: Johnston FE, Foster GD (Eds.) Obesity, Growth and Development. London, UK: Smith-Gordon and Company Limited Publishers, 2001, pp.129-141.